CLINICAL TRIAL: NCT03038737
Title: Comparative Study Of Biting Force Of Injection Molded PEEK and Bre.Flex Materials For Bounded Removable Partial Dentures (Randomized Clinical Trial)
Brief Title: Comparative Study of Biting Force of Injection Molded PEEK and Bre.Flex for Removable Partial Dentures.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Arwa Mabrouk Ayad Issa, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 1234
Record Dates: First submitted 2017-01-26; First posted 2017-02-01 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Biting
Keywords: nylon; polyamide; PEEK; partial denture
MeSH Terms: conditions — Bites and Stings | interventions — polyetheretherketone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Active Comparator): patients will receive partial denture constructed from breflex material
  Interventions: Other: bre.flex
- group 2 (Experimental): patients will receive partial denture constructed from PEEK material
  Interventions: Other: PEEK

INTERVENTIONS:
Other: bre.flex — In the recent time thermoplastic materials become quite popular in clinical practice such as nylon and acetal resins. since the 1950, polyamide resin (nylons) provide improved esthetics and reduction of rotational forces on the abutment teeth due to their low elastic modulus(3).
  The major disadvantage of a nylon RDP is the inability for a reline procedure and the lack of occlusal rests as well as rigid frameworks, that could lead to occlusal instability and sinking, especially in Kennedy class I and II cases. On the other hand, acetal resins present adequate mechanical strength to form a frame-work more rigid than nylon with retentive clasps, connectors, and supportive elements; however, the acetal resin material lacks natural translucency and vitality.
  Arms: group 1
Other: PEEK — PEEK has been successfully used over the last years in the medical ﬁeld, and orthopedics, speciﬁcally. which presents high biocompatibility, good mechanical properties, high temperature resistance, and chemical stability due to a 4 GPa modulus of elasticity, it is as elastic as bone and can reduce stresses transferred to the abutment teeth.Additional advantages of this polymer material are elimination of allergic reactions and metallic taste, high polishing qualities, low plaque afﬁnity, and good wear resistance, it has only recently been used in dentistry.
  Arms: group 2

SUMMARY:
The aim of the present study is to evaluate the biting force of upper removable partial denture constructed from two different flexible thermoplastic materials.

DETAILED DESCRIPTION:
The patient will be treated in visits designated as follows:

Visit 1: Preoperative records, clinical, radiographic examination (panoramic and periapical x-rays for evaluation the crown-root ratio, the apical condition of the abutment and their alveolar bone support of abutment) and primary impression will be performed with irreversible hydro-colloid impression material (alginate), The impressions will be poured with type IV dental stone to obtain diagnostic casts .

Visit 2: Maxillary Face-bow will be recorded. The diagnostic casts will be mounted on semi adjustable articulator in centric occluding relation to evaluate the interarch distance and occlusal plane.

Visit 3: primary surveying is performed. Special trays will be constructed and Mouth preparation will be performed by preparing guiding planes and rests seats will be prepared opposing to the edentulous area. Final impression will be taken by elastomeric impression material. The impression will be poured into type IV dental stone in order to obtain master cast. The master cast will be surveyed. The proposed design will be as follows: metal framework base saddle for edentulous areas on both sides connected with palatal strap. Aker's clasp on all abutments with buccal retention.

Visit 4: the metal framework is tried into the patient's mouth. Jaw relation is recorded.

Visit 5: The denture base will be tried in with acrylic teeth in patient's mouth.

Visit 6: the denture base of the partial denture will be processed incorporation with the metal framework into the two different materials to be evaluated. The first group will receive the partial denture in which the metal framework incorporated with the denture base fabricated from PEEK material. The second group will receive the partial denture in which the metal framework incorporated with the denture base material fabricated from BRE-FLEX.

Visit7,8,9: clinical measurement will be performed for one month in three visits.

ELIGIBILITY:
Inclusion Criteria:

* i. All patients must have Kennedy class III modification I upper partially edentulous ridges.

ii. The remaining teeth have good periodontal condition, with no signs of attrition or gingival recession.

iii. Male or female patient with age range (45-55) and in good medical condition iv. All patients have skeletal Angle's class I maxillo-mandibular relationship and have sufficient interarch distance.

v. Free from any systemic or neuromuscular disorder that might affect chewing efficiency of masticatory muscles.

vi. Free from any tempro-mandibular joint disorder. vii. The patients have good oral hygiene and low caries index.

Exclusion Criteria:

* i. Patients having abnormal habits as bruxism or clenching ii. Patients having hormonal disorders as diabetes, thyroid or parathyroid hormonal diseases were not included.

iii. Teeth with compromised bone support. iv. Patient with xerostomia or excessive salivation. v. Patient with abnormal tongue behavior and/or size.

Ages: 45 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-03 (Estimated); Primary Completion 2017-08 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
change in Biting force | 1 month
  the change in biting force will be recorded three times. The first week at the time of insertion measuring the biting force immediately after partial denture insertion. The third week measuring biting force of the partial denture. The fourth week measuring biting force of the partial denture.
  the biting force will be measured by I-load sensor.

IPD SHARING:
Plan to Share IPD: Undecided